CLINICAL TRIAL: NCT01706991
Title: MEPEDS New Device Pediatric Vision Scanner
Brief Title: Amblyopia and Strabismus Detection Using a Pediatric Vision Scanner
Status: Completed | Type: Observational
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: rebiscan-003
Record Dates: First submitted 2012-10-05; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Amblyopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Normal Controls: Structurally normal eye with equal visual acuity and normal stereopsis.
  Interventions: Device: Pediatric Vision Scanner eye scan
- Referral required: Diagnosed with amblyopia or constant strabismus, categorized based on the GSE.
  Amblyopia:
  * VA <20/40 and 2 logMAR lines difference in normal eye
  * Mild amblyopia (>20/40)
  * Moderate amblyopia (20/40 and <20/100)
  * Severe amblyopia (≥20/100 or worse)
  * Bilateral amblyopia: >4 years age VA<20/40 OU including high hyperopia or high astigmatism.
  Strabismus:
  * Constant: >2 PD at near and or distance.
  * Intermittent: strabismus that could be controlled intermittently either through fusional mechanisms or a compensatory head position.
  Amblyogenic factor categorization:
  * 'Anisometropia'- (1.5 Diopters (D) or more difference in refractive error between the two eyes.
  * 'hypermetropia' (≥3.5 D),
  * 'myopia' (≥-4.0 D),
  * 'astigmatism' (≥1.5 D).
  * 'structural abnormalities' of the eye will not be excluded, but will be considered to have vision loss if visual acuity is 20/40 or worse.
  Interventions: Device: Pediatric Vision Scanner eye scan
- Borderline: (no long-term harm to patient if referral is delayed, however the patient does have conditions that might benefit from monitoring): Equal visual acuity and no structural abnormality with any of the following: Amblyogenic factor, intermittent strabismus, structural abnormalities, refractive error, reduced stereopsis.
  Interventions: Device: Pediatric Vision Scanner eye scan

INTERVENTIONS:
Device: Pediatric Vision Scanner eye scan — Subject is scanned with a 2.5 second pediatric vision scanner device test.

SUMMARY:
The purpose of this project is to compare the performance of the Pediatric Vision Scanner (PVS) with the Gold Standard Examination to determine the effectiveness of the PVS at detecting amblyopia and strabismus. All tests and observations will be done at a single visit over the course of approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 6 years
* Signed Informed consent by parent or guardian
* Meet all inclusion criteria.

Exclusion Criteria:

* Children with a history of developmental delay or cognitive deficit
* Children unable to complete the GSE (including visual acuity testing)

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children presenting for ophthalmic exam at eye clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Binocularity score | Day 1

SECONDARY OUTCOMES:
Presence of amblyopia risk factors | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Varma, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- Doheny Eye Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Loudon SE, Rook CA, Nassif DS, Piskun NV, Hunter DG. Rapid, high-accuracy detection of strabismus and amblyopia using the pediatric vision scanner. Invest Ophthalmol Vis Sci. 2011 Jul 7;52(8):5043-8. doi: 10.1167/iovs.11-7503. PMID 21642624